CLINICAL TRIAL: NCT01522924
Title: Tobacco Dependence Treatment Education for Dental Students Using Standardized Patients
Brief Title: Tobacco Dependence Treatment Education for Dental Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Jacqueline A. Singleton, Associate Professor, University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12.0026
Record Dates: First submitted 2012-01-24; First posted 2012-02-01 (Estimated); Results first posted 2013-08-22 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Smoking
Keywords: tobacco cessation treatment; standardized patients; dental students; tobacco cessation treatment education
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counseling practice sessions (Experimental): Dental students will be administered the first questionnaire before receiving a tobacco cessation lecture and the second questionnaire after the lecture, counseling practice sessions using standardized patients, and debriefing session.
  Interventions: Other: Counseling practice sessions
- Lecture only (No Intervention): Students will receive the first questionnaire before the lecture and the second questionnaire after the lecture

INTERVENTIONS:
Other: Counseling practice sessions — Dental students will complete the first questionnaire before a tobacco cessation lecture and the second questionnaire after the lecture, counseling practice sessions using standardized patients and a debriefing session.
  Other Names: Tobacco cessation treatment education; Tobacco cessation counseling; Smoking cessation counseling; Tobacco dependence treatment; Standardized patients
  Arms: Counseling practice sessions

SUMMARY:
This study determines if there is a difference in dental students' attitudes, perceived barriers, subjective norms, perceived skills, self-efficacy, intentions to provide cessation treatment, and cessation knowledge in those students receiving a tobacco cessation lecture along with practice sessions using standardized patients and those students receiving only a tobacco cessation lecture. The study determines if dental students' use of tobacco affects their intent to provide cessation treatment to patients, and if the time between receiving the lecture and participating in the practice sessions using standardized patients makes a difference in dental students' attitudes, perceived barriers, subjective norms. perceived skills, self-efficacy, intentions to provide cessation treatment, and cessation knowledge.

DETAILED DESCRIPTION:
The experimental study has a pretest-posttest design. It evaluates the changes to dental students' attitudes, perceived barriers, subjective norms, perceived skills, self-efficacy, intentions to provide cessation treatment, and tobacco cessation knowledge between those students receiving a lecture along with practice sessions using standardized patients and those students receiving only a lecture. Dental students will be invited to complete two questionnaires. The control group of dental students will complete the first questionnaire before the lecture and the second questionnaire after the lecture. The experimental group of dental students will complete the first questionnaire before the lecture and the second questionnaire after the lecture and the practice and debriefing sessions. Subjects will include 120 first year dental students in an introductory course to clinical dentistry. The cessation training is a required activity in the course. Students are divided into small groups according to their bench or lab numbers. These numbers are assigned to the student based on the alphabetical order of their name. The eligibility criteria is: 1) Must be a first year dental student in Introduction to Clinical Dentistry 1 at the University of Louisville, and 2) Must be willing to volunteer to complete pre- and post-questionnaires about the cessation treatment educational program. The exclusion criteria is: Subject is not willing to give consent to complete the pre- and post- questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* must be a first year dental student in Introduction to Clinical Dentistry I at the study institution
* volunteer to complete pre- and post-questionnaires concerning tobacco cessation treatment educational training.

Exclusion Criteria:

* subject does not complete pre- and post- questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline A Singleton, MEd, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville School of Dentistry, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Walsh SE, Singleton JA, Worth CT, Krugler J, Moore R, Wesley GC, Mitchell CK. Tobacco cessation counseling training with standardized patients. J Dent Educ. 2007 Sep;71(9):1171-8. PMID 17761623
- See also: Centers for Disease Control and Prevention — http://www.cdc.gov/tobacco
- See also: American Cancer Society — http://www.cancer.org
- See also: American Dental Association — http://www.ada.org
- See also: American Dental Hygienists' Association — http://www.adha.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period began on February 23 and ended on April 19. The location of the study was at a dental school and the standardized patient clinic in the medical school.
Pre-assignment Details: Students were excluded from the study if they did not meet study requirements.
Period: Overall Study
Arm/Group | Counseling Practice Sessions | Lecture Only
Started | 42 (There were 42 dental students in the intervention group.) | 52 (There were 52 dental students in the control group.)
Completed | 42 (There were 42 dental students who completed the second survey after the intervention.) | 52 (There were 52 dental students who completed the second survey after the lecture.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 94 dental students who provided linkable surveys. There were 42 in the intervention group and 52 in the control group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Counseling Practice Sessions | Lecture Only | Total
Number analyzed (Participants) | 42 | 52 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 52 | 94
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.66 (4.31) | 25.00 (3.74) | 25.29 (3.99)
Sex/Gender, Customized [Number; unit: participants] — Missing data on one participant. Data is unknown.
  participants
    Female | 12 | 23 | 35
    Male | 29 | 29 | 58
Region of Enrollment [Number; unit: participants]
  United States | 42 | 52 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attitude Score
Description: The attitude variable was computed by adding the values from two questionnaire items to assess the level agreement with statements: 1.) "It is important for members of the profession to discuss tobacco use with patients" and 2.) "A brief intervention (3 minutes) for tobacco cessation with my patients would be effective." The rating scale was: 0 = strongly disagree, 1 = moderately disagree, 2 = somewhat disagree, 3 = neither disagree or agree, 4 = somewhat agree, 5 = moderately agree, and 6 = strongly agree. A higher value represents participants' more positive attitude toward providing tobacco cessation treatment (Range:0-8). The difference in the attitude from Questionnaire 1 to Questionnaire 2 was computed by subtracting the total value of the variable at Questionnaire 1 from the total value at Questionnaire 2.
Time Frame: Questionnaire 1 (baseline/pre-lecture) to Questionnaire 2 (post-lecture or post-lecture and counseling/debriefing sessions)
Population: The control group (lecture only) completed the second questionnaire after the lecture and the intervention group (counseling practice sessions) completed the second questionnaire after the counseling practice sessions and the debriefing session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Counseling Practice Sessions | Lecture Only
Number analyzed (Participants) | 42 | 52
units on a scale | .64 (2.61) | -.25 (2.27)

2. Primary Outcome: Change From Baseline in Perceived Barriers Score
Description: The perceived barriers variable was computed by adding the total number of barriers reported by participants. Participants were asked to select all factors that may limit their ability to counsel tobacco users during every visit. The rating scale for reporting barriers was: 0 = no and 1 = yes. A higher value represents a higher number of barriers to providing tobacco cessation treatment reported by participants(Range: 0-11). The difference in perceived barriers from Questionnaire 1 to Questionnaire 2 was computed by subtracting the total number of perceived barriers at Questionnaire 1 from the total number of perceived barriers at Questionnaire 2.
Time Frame: Questionnaire 1(baseline/pre-lecture) to Questionnaire 2(post-lecture or post-lecture and counseling /debriefing sessions)
Population: The number of participants for analysis was determined by completing the second questionnaire after the lecture or after the counseling practice sessions using standardized patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Counseling Practice Sessions | Lecture Only
Number analyzed (Participants) | 42 | 52
units on a scale | 1.83 (1.53) | .87 (1.78)

3. Primary Outcome: Change From Baseline in Subjective Norms Score
Description: Subjective norms are beliefs that people who influence your actions approve or disapprove of the behavior. The subjective norms variable was computed by adding the values of six questions to assess the participants' level of perceived social pressures to counsel patients in quitting tobacco use. Questions wer rated on a seven-point Likert scale; higher point values indicate a perceived social norm more supportive of counseling patients in quitting tobacco use(Range: 0-36). The difference in the subjective norms score from Questionnaire 1 to Questionnaire 2 was computed by subtracting the total number of participants' subjective norms at Questionnaire 1 from the total number of participants' subjective norms at Questionnaire 2.
Time Frame: Questionnaire 1 ( baseline/pre-lecture) to Questionnaire 2 (post-lecture or post-lecture and counseling/debriefing sessions)
Population: The number of participants for analysis was determined by the completing the questionnaire after the lecture or after the counseling practice sessions using standardized patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Counseling Practice Sessions | Lecture Only
Number analyzed (Participants) | 42 | 52
units on a scale | 2.55 (4.73) | .67 (3.42)

4. Primary Outcome: Change From Baseline in Perceived Skills Score
Description: The perceived skills variable was computed by adding the values of seven questions that assessed the participants' perceived level of tobacco cessation treatment skills from poor to excellent. The rating scale was: 0 = poor, 1 = fair, 2 = good, 3 = very good, and 4 = excellent. A higher value represents a higher level of tobacco cessation treatment skills perceived by participants (Range: 0-28). The difference in the participants' perceived skills from Questionnaire 1 to Questionnaire 2 was computed by subtracting the total value of perceived skills at Questionnaire 1 from the total value of perceived skills at Questionnaire 2.
Time Frame: Questionnaire 1(baseline/pre-lecture) to Questionnaire 2 (post-lecture or post-lecture and counseling/debriefing sessions)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Counseling Practice Sessions | Lecture Only
Number analyzed (Participants) | 42 | 52
units on a scale | 8.52 (6.62) | 3.38 (4.84)

5. Primary Outcome: Change From Baseline in Self-efficacy Score
Description: Self-efficacy represents an individual's confidence in his/her ability to perform a behavior. The self-efficacy variable was computed by adding the values of ten questions to assess the participants' self-efficacy to counsel patients to quit tobacco use. The rating scale was: 0 = not at all confident, 1 = not very confident, 2 = moderately confident, 3 = very confident, and 4 = extremely confident. A higher value represents participants' higher level of confidence in providing tobacco cessation treatment (Range: 0-40). The difference in participants' self-efficacy from Questionnaire 1 to Questionnaire 2 was computed by subtracting the total value of self-efficacy at Questionnaire 1 from the total value at Questionnaire 2.
Time Frame: Questionaire 1 (baseline/pre-lecture) to Questionnaire 2 (post-lecture or post-lecture and counseling/debriefing sessions)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Counseling Practice Sessions | Lecture Only
Number analyzed (Participants) | 42 | 52
units on a scale | 14.34 (8.61) | 7.66 (6.90)

6. Primary Outcome: Change From Baseline in Intentions Score
Description: Participants' intentions to provide tobacco cessation treatment were computed by adding values from thirteen questions to assess dental students' intent to counsel patients to quit tobacco use. The rating scale was: 0 = never, 1 = rarely, 2 = sometimes, 3 = almost always, 4 = always (every visit). A higher value represents participants' stronger intentions to provide tobacco cessation treatment (Range: 0-52). The difference in participants' intentions to provide tobacco cessation treatment from Questionnaire 1 to Questionnaire 2 was computed by subtracting the total value of participants' intentions at Questionnaire 1 from the total value of participants' intentions at Questionnaire 2.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Counseling Practice Sessions | Lecture Only
Number analyzed (Participants) | 42 | 52
units on a scale | 7.88 (9.05) | 1.90 (6.96)

7. Primary Outcome: Change From Baseline in Tobacco Cessation Knowledge Score
Description: The tobacco cessation knowledge variable was computed by adding the participants' total number of correct answers of the ten knowledge questions. The rating scale was: 0 = incorrect and 1 = correct. A higher value represents participants' higher level of tobacco cessation treatment knowledge (Range: 0-10). The difference in the tobacco cessation knowledge from Questionnaire 1 to Questionnaire 2 was computed by subtracting the total number of participants' correct answers at Questionnaire 1 from the total number of participants' correct answers at Questionnaire 2.
Time Frame: Questionnaire 1 (pre-lecture) to Questionnaire 2 (post-lecture or post-lecture and counseling/debriefing sessions)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Counseling Practice Sessions | Lecture Only
Number analyzed (Participants) | 42 | 52
units on a scale | 2.55 (2.98) | 2.60 (2.77)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Serious and nonserious adverse events were not collected for either arm of the study.
Groups:
- Lecture Only: participated in lecture only
- Counseling/Debriefing: participated in counseling and debriefing sessions
Arm/Group | Lecture Only | Counseling/Debriefing
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
One participant in the intervention group did not provide gender information. The total number of participants in the intervention group did not equal the number of male and female participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes